CLINICAL TRIAL: NCT05947500
Title: A Randomized Phase 2 Study of ATR Inhibition in Advanced PD-(L)1-Refractory Merkel Cell Carcinoma: The MATRiX Trial
Brief Title: Testing the Combination of Two Anticancer Drugs M1774 (Tuvusertib) and Avelumab to Evaluate Their Safety and Effectiveness in Treating Merkel Cell Skin Cancer, MATRiX Trial
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2023-05259; NCI-2023-05259 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10592 (Other: Dana-Farber - Harvard Cancer Center LAO); 10592 (Other: CTEP); P30CA015704 (NIH)
Record Dates: First submitted 2023-07-13; First posted 2023-07-17 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-10

CONDITIONS: Clinical Stage III Cutaneous Merkel Cell Carcinoma AJCC v8; Clinical Stage IV Cutaneous Merkel Cell Carcinoma AJCC v8; Locally Advanced Merkel Cell Carcinoma; Metastatic Merkel Cell Carcinoma; Refractory Merkel Cell Carcinoma; Unresectable Merkel Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Merkel Cell | interventions — avelumab; Biopsy; Specimen Handling; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (tuvusertib) (Active Comparator): Patients receive tuvusertib PO QD on days 1-14 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT, PET/CT, or MRI, biopsy, and collection of blood and stool at screening and on study. Patients with documented progression may cross over to Arm 2. (CLOSED TO ACCRUAL 5/12/2025)
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Drug: Tuvusertib
- Arm 2 (tuvusertib, avelumab) (Experimental): Patients receive tuvusertib PO QD on days 1-14 of each cycle and avelumab IV over 60 minutes on day 1 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT, PET/CT, or MRI, biopsy, and collection of blood and stool at screening and on study.
  Interventions: Drug: Avelumab; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Drug: Tuvusertib

INTERVENTIONS:
Drug: Avelumab — Given IV
  Other Names: Bavencio; MSB 0010718C; MSB-0010718C; MSB0010718C
  Arms: Arm 2 (tuvusertib, avelumab)
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood and stool
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Drug: Tuvusertib — Given PO
  Other Names: ATR Kinase Inhibitor M1774; M 1774; M-1774; M1774

SUMMARY:
This phase II trial compares tuvusertib in combination with avelumab to tuvusertib alone to determine whether the combination therapy will lengthen the time before the cancer starts getting worse in patients with Merkel cell cancer that has not responded to previous treatment (refractory). Tuvusertib is a drug that inhibits an enzyme called ataxia telangiectasia and Rad3 related (ATR) kinase, which is an enzyme that plays a role in repair of damaged deoxyribonucleic acid (DNA) as well as tumor cell replication and survival. It may lead to tumor cell death by inhibiting ATR kinase activity. Immunotherapy with monoclonal antibodies, such as avelumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving tuvusertib in combination with avelumab may lengthen the time before Merkel cell cancer starts getting worse compared to giving avelumab alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the potential efficacy, using progression free survival (PFS), of ATR inhibition alone to ATR inhibition plus anti-PD-(L)1 therapy through a randomized clinical trial for patients with advanced Merkel cell carcinoma (MCC) who have progressed on anti-PD(L)1 therapy.

SECONDARY OBJECTIVES:

I. To compare the clinical activity of ATR inhibition alone to that in combination with avelumab through a randomized clinical trial for patients with advanced MCC that has progressed after PD-1 pathway blockade.

II. To identify gene expression-based immunologic (replication stress / neuroendocrine [NE] differentiation) signatures predictive of response to ATR inhibition in advanced immunotherapy-refractory MCC tumors through ribonucleic acid sequencing (RNAseq).

EXPLORATORY OBJECTIVES:

I. To examine the association of various biomarkers with the clinical activity of ATR inhibition alone or in combination with PD-(L)1 pathway blockade.

II. To explore the safety and efficacy (PFS, overall response rate [ORR], and overall survival [OS]) of the addition of avelumab to M1774 (tuvusertib) after documented progressive disease of M1774 (tuvusertib) monotherapy.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM 1 (CLOSED TO ACCRUAL 5/12/2025): Patients receive tuvusertib orally (PO) once daily (QD) on days 1-14 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT), positron emission tomography (PET)/CT, or magnetic resonance imaging (MRI), biopsy, and collection of blood and stool/rectal swabs at screening and on study. Patients with documented progression may cross over to Arm 2.

ARM 2: Patients receive tuvusertib PO QD on days 1-14 of each cycle and avelumab intravenously (IV) over 60 minutes on day 1 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT, PET/CT, or MRI, biopsy, and collection of blood and stool at screening and on study.

After completion of study treatment, patients are followed up at 30 days and then every 6 months for 2 years from the last dose of treatment.

ELIGIBILITY:
Inclusion Criteria:

* REGISTRATION ELIGIBILITY: Patients must have a history of pathologically confirmed locally advanced/unresectable Merkel cell carcinoma or metastatic Merkel cell carcinoma
* REGISTRATION ELIGIBILITY: Patients must have evaluable disease per Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1
* REGISTRATION ELIGIBILITY: Patients must have had prior treatment with anti-PD-1 or anti-PD-L-1 antibody (e.g., pembrolizumab, avelumab, etc.) and have experienced progressive disease during treatment or within 120 days from the last dose of anti-PD-(L)1 therapy. Anti-PD-(L)1 therapy administered in combination with other agent(s) including ipilimumab is also allowed as prior therapy, if patients experienced progressive disease during treatment or within 120 days from the last dose of anti-PD-(L)1 therapy. The last dose of anti-PD-(L)1 antibody must be ≥ 14 days prior to planned C1D1. If participants are receiving or received cytotoxic chemotherapy as most recent therapy prior to screening for this trial, there must be clinically and/or radiologically documented progressive disease on or after chemotherapy prior to being eligible for this study. If the patient is receiving bridging chemotherapy, the most recent administration must be ≥ 14 days prior to planned cycle 1 day 1 (C1D1) of the clinical trial to be eligible
* REGISTRATION ELIGIBILITY: Age >= 18 years. Because no dosing or adverse event data are currently available on the use of M1774/tuvusertib in combination with avelumab in patients < 18 years of age, children are excluded from this study
* REGISTRATION ELIGIBILITY: Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* REGISTRATION ELIGIBILITY: Absolute neutrophil count >= 1,000/mcL
* REGISTRATION ELIGIBILITY: Platelets >= 100,000/mcL
* REGISTRATION ELIGIBILITY: Total bilirubin =< institutional upper limit of normal (ULN) or ≤ 1.5 x ULN for subjects with Gilbert's disease
* REGISTRATION ELIGIBILITY: Aspartate aminotransferase (AST)(serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x institutional ULN
* REGISTRATION ELIGIBILITY: Serum creatinine =< 1.5 x institutional ULN

  * (If serum creatinine is > 1.5 x ULN, creatinine clearance needs to be ≥ 50 mL/min by Cockcroft-Gault calculation or by a measured 24-hour urine collection for the participant to be eligible.)
* REGISTRATION ELIGIBILITY: Hemoglobin >= 9.0 g/dL
* REGISTRATION ELIGIBILITY: Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* REGISTRATION ELIGIBILITY: For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* REGISTRATION ELIGIBILITY: Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* REGISTRATION ELIGIBILITY: Patients with treated brain metastases are eligible if follow-up brain imaging during screening shows no evidence of progressive brain metastases and it has been at least 4 weeks since central nervous system (CNS) directed therapy
* REGISTRATION ELIGIBILITY: Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* REGISTRATION ELIGIBILITY: Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* REGISTRATION ELIGIBILITY: The effects of M1774(tuvusertib) on the developing human fetus are unknown. For this reason and because ATR inhibitor agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and, for the duration of study participation, and 6 months after completion of M1774 (tuvusertib) and avelumab administration. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 3 months after completion of M1774 (tuvusertib) and avelumab administration
* REGISTRATION ELIGIBILITY: Ability to understand and the willingness to sign a written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants
* CROSSOVER ELIGIBILITY: Patient was initially assigned to arm 1 (M1774/tuvusertib monotherapy) and completed at least 21 of 28 possible doses of M1774/ tuvusertib
* CROSSOVER ELIGIBILITY: Patients must have documented progressive disease per RECIST v 1.1
* CROSSOVER ELIGIBILITY: ECOG performance status ≤ 2 (Karnofsky ≥ 60%)
* CROSSOVER ELIGIBILITY: Absolute neutrophil count ≥ 1,000/mcL (within 14 days of crossover registration)
* CROSSOVER ELIGIBILITY: Platelets ≥ 100,000/mcL (within 14 days of crossover registration)
* CROSSOVER ELIGIBILITY: Total bilirubin ≤ institutional upper limit of normal (ULN) or ≤ 1.5 x ULN for subjects with Gilbert's disease (within 14 days of crossover registration)
* CROSSOVER ELIGIBILITY: AST(SGOT)/ALT(SGPT) ≤ 3 × institutional ULN (within 14 days of crossover registration)
* CROSSOVER ELIGIBILITY: Serum creatinine ≤ 1.5 x institutional ULN (within 14 days of crossover registration)

  * (If serum creatinine is > 1.5 x ULN, creatinine clearance needs to be ≥ 50 mL/min by Cockcroft-Gault calculation or by a measured 24-hour urine collection for the participant to be eligible.)
* CROSSOVER ELIGIBILITY: Hemoglobin ≥ 9.0 g/dL (within 14 days of crossover registration)
* CROSSOVER ELIGIBILITY: Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* CROSSOVER ELIGIBILITY: For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* CROSSOVER ELIGIBILITY: Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* CROSSOVER ELIGIBILITY: Patients with treated brain metastases are eligible if follow-up brain imaging during screening shows no evidence of progressive brain metastases and it has been at least 4 weeks since central nervous system (CNS) directed therapy
* CROSSOVER ELIGIBILITY: Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* CROSSOVER ELIGIBILITY: Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* CROSSOVER ELIGIBILITY: The effects of M1774 (tuvusertib) on the developing human fetus are unknown. For this reason and because ATR inhibitor agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and, for the duration of study participation, and 6 months after completion of M1774 (tuvusertib) and avelumab administration. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 3 months after completion of M1774 (tuvusertib) and avelumab administration

Exclusion Criteria:

* REGISTRATION EXCLUSION: Patients with life-threatening immune-related adverse events (IRAEs) related to prior anti-PD-(L)1 antibody. Patients with a history of IRAE of grade 4 (G4) severity (excluding thyroid or endocrine disorders now controlled) or IRAE of any severity that required permanent treatment discontinuation with prior immune checkpoint inhibitor (ICI) therapy due to toxicity
* REGISTRATION EXCLUSION: Patients with a prior history of ataxia telangiectasia
* REGISTRATION EXCLUSION: Patients who are receiving any other investigational agents
* REGISTRATION EXCLUSION: History of allergic reactions attributed to compounds of similar chemical or biologic composition to M1774/tuvusertib or avelumab
* REGISTRATION EXCLUSION: Patients with uncontrolled intercurrent illness or any other significant condition(s) that would make participation in this protocol unreasonably hazardous
* REGISTRATION EXCLUSION: Pregnant women are excluded from this study because M1774 (tuvusertib) and avelumab have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with M1774 (tuvusertib) and avelumab breastfeeding should be discontinued if the mother is treated with M1774 (tuvusertib) or avelumab and for at least 1 month after the last dose of study medications. These potential risks may also apply to other agents used in this study
* REGISTRATION EXCLUSION: Patients who are not able to swallow orally administered medication or have gastrointestinal disorders likely to interfere with absorption of the study medication
* REGISTRATION EXCLUSION: Patients who cannot discontinue proton-pump inhibitors (PPIs)
* REGISTRATION EXCLUSION: Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia and neuropathy, which may be =< grade 2. Patients with endocrinopathies requiring hormone replacement (such as hypothyroidism, autoimmune diabetes mellitus, adrenal insufficiency) will be allowed
* REGISTRATION EXCLUSION: M1774/ tuvusertib is primarily metabolized by aldehyde oxidase and to a lesser extent CYP3A4 and CYP1A2; therefore, concomitant administration with strong inhibitors of CYP3A4 (e.g., ketoconazole, itraconazole, clarithromycin, ritonavir, indinavir, nelfinavir and saquinavir) and CYP1A2 or inducers of CYP3A4 (e.g. rifampin, phenytoin, carbamazepine, phenobarbital, St. John's Wort) and CYP1A2 are prohibited. M1774/ tuvusertib is an inhibitor of MATE1 and MATE2K and substrates of these transporters are also prohibited. These include metformin, acyclovir, estrone sulfate, ciprofloxacin and cephalexin. Patients who are taking such medications who cannot discontinue or switch them to an acceptable alternative are not eligible

  * Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference for a list of drugs to avoid or minimize use of. One example of such a reference is here (https://go.drugbank.com/categories/DBCAT003956)
  * As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* REGISTRATION EXCLUSION: Patients who are on chronic corticosteroid treatment exceeding 10 mg prednisone daily (or equivalent) are excluded. Chronic corticosteroid use lower than this range is permitted
* REGISTRATION EXCLUSION: Patients with a QTcF (using the Fridericia correction calculation) of > 470 msec
* CROSSOVER EXCLUSION: Patients with life-threatening immune-related adverse events (IRAEs) related to prior anti-PD-(L)1 antibody. Patients with a history of IRAE of G4 severity (excluding thyroid or endocrine disorders now controlled) or IRAE of any severity that required permanent treatment discontinuation with prior ICI therapy due to toxicity
* CROSSOVER EXCLUSION: Patients with a prior history of ataxia telangiectasia.
* CROSSOVER EXCLUSION: Patients who are receiving any other investigational agents
* CROSSOVER EXCLUSION: History of allergic reactions attributed to compounds of similar chemical or biologic composition to M1774/tuvusertib or avelumab
* CROSSOVER EXCLUSION: Patients with uncontrolled intercurrent illness or any other significant condition(s) that would make participation in this protocol unreasonably hazardous
* CROSSOVER EXCLUSION: Pregnant women are excluded from this study because M1774 (tuvusertib) and avelumab have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with M1774 (tuvusertib) and avelumab breastfeeding should be discontinued if the mother is treated with M1774 (tuvusertib) or avelumab and for at least 1 month after the last dose of study medications. These potential risks may also apply to other agents used in this study
* CROSSOVER EXCLUSION: Patients who are not able to swallow orally administered medication or have gastrointestinal disorders likely to interfere with absorption of the study medication
* CROSSOVER EXCLUSION: Patients who cannot discontinue proton-pump inhibitors (PPIs)
* CROSSOVER EXCLUSION: Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia and neuropathy which may be ≤ grade 2. Additionally, anemia felt related to M1774/tuvusertib may be grade 2 as long as it exceeds requirement of hemoglobin > 9 g/dL. Patients with endocrinopathies requiring hormone replacement (such as hypothyroidism, autoimmune diabetes mellitus, adrenal insufficiency) will be allowed
* CROSSOVER EXCLUSION: M1774/ tuvusertib is primarily metabolized by aldehyde oxidase and to a lesser extent CYP3A4 and CYP1A2; therefore, concomitant administration with strong inhibitors of CYP3A4 (e.g., ketoconazole, itraconazole, clarithromycin, ritonavir, indinavir, nelfinavir and saquinavir) and CYP1A2 or inducers of CYP3A4 (e.g. rifampin, phenytoin, carbamazepine, phenobarbital, St. John's Wort) and CYP1A2 are prohibited. M1774/ tuvusertib is an inhibitor of MATE1 and MATE2K and substrates of these transporters are also prohibited. These include metformin, acyclovir, estrone sulfate, ciprofloxacin and cephalexin. Patients who are taking such medications who cannot discontinue or switch them to an acceptable alternative are not eligible. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference for a list of drugs to avoid or minimize use of. One example of such a reference is here (https://go.drugbank.com/categories/DBCAT003956). Patient Drug Information Handout and Wallet Card) should be provided to patients. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* CROSSOVER EXCLUSION: Patients who are on chronic corticosteroid treatment exceeding 10 mg prednisone daily (or equivalent) are excluded. Chronic corticosteroid use lower than this range is permitted
* CROSSOVER EXCLUSION: Patients with a QTcF (using the Fridericia correction calculation) of > 470 msec

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-05-21 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Composite progression-free survival (PFS) | From registration to progressive disease or death whichever occurs first, assessed up to 2 years
  The stratified (on disease, acquired versus primary immune checkpoint inhibitor-refractory disease) log-rank test will be used to compare PFS between arms. The primary analysis will be done on an intent-to-treat basis. An as-treated analysis will also be done as a sensitivity analysis.

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 2 years
  The sum of complete and partial responses per Response Evaluation Criteria in Solid Tumors 1.1 criteria. Evaluated using the Mantel-Haenszel test.
Duration of response | From the time measurement criteria are met for complete or partial response (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented, assessed up to 2 years
  Will be evaluated by estimating the probability of response using a cumulative incidence estimate, and then among those who responded, creating a time-to-recurrence curve using a cumulative-incidence estimate. Will be compared between arms using the stratified log-rank test and the Mantel-Haenszel test will be used to compare binary outcomes.
Overall survival (OS) | Up to 2 years
  Will be evaluated using a stratified log-rank test. Will be compared between arms using the stratified log-rank test and the Mantel-Haenszel test will be used to compare binary outcomes.
Gene expression-based immunologic signatures predictive of response | Up to 2 years
  Annotated transcriptome sequences at baseline and on-therapy will be correlated with response in both virus-positive and -negative tumors. Descriptive statistical analyses will be performed. Volcano plots will be evaluated. Gene set enrichment analysis will be used to compare pre-treatment samples from patients with response to treatment to samples from patients experiencing disease progression. The Kolmogorov-Smirnov test will be used to test for statistical differences followed by the Bonferroni correction to adjust for multiple comparisons.

OTHER OUTCOMES:
Biomarker levels | Up to 2 years
  Will examine the association of various biomarkers with the primary and secondary endpoints. All patients will be combined for these purposes, and separate examination of biomarkers will be conducted by treatment group to allow for the possibility that certain correlates will have differing associations with outcome according to treatment group. This will be done using logistic regression for ORR and Cox regression for OS and PFS. In addition, descriptive statistics for biomarkers will be presented (mean, standard deviation, median, and interquartile range) by treatment group and based on presence or absence of response. Biomarker levels will also be compared between the two treatment groups using the two-sample t-test (or the non-parametric Wilcoxon rank-sum test as needed).

CONTACTS AND LOCATIONS:
Overall Officials: Paul Nghiem, Principal Investigator — Fred Hutchinson Cancer Center
Locations (51):
- United States (50):
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Keck Medicine of USC Koreatown, Los Angeles, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - UM Sylvester Comprehensive Cancer Center at Aventura, Aventura, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Moffitt Cancer Center - McKinley Campus, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Memorial Hospital East, Shiloh, Illinois
  - HaysMed, Hays, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Hospital-Indian Creek Campus, Overland Park, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington
- University Health Network-Princess Margaret Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

DOCUMENTS (1):
  • Informed Consent Form (2025-08-04): https://cdn.clinicaltrials.gov/large-docs/00/NCT05947500/ICF_000.pdf